CLINICAL TRIAL: NCT06286475
Title: A Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of VRG50635 in Healthy Volunteers
Brief Title: A Study of VRG50635 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verge Genomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VGCS-50635-003
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Amyotrophic lateral sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a 2-part study that includes both an open-label (Part 1) and a double-blind, placebo-controlled (Part 2) design. In Part 1, participants will be randomly assigned to receive open-label VRG50635 in 1 of 2 treatment sequences. In Part 2, participants will receive VRG50635 or placebo in a double-blind manner.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: VRG50635 Sequence A, B, C (Experimental): Participants will receive a single dose of VRG50635 in each of 3 treatment periods separated by 14-day washout periods.
  Interventions: Drug: VRG50635
- Part 1: VRG50635 Sequence B, A, C (Experimental): Participants will receive a single dose of VRG50635 in each of 3 treatment periods separated by 14-day washout periods.
  Interventions: Drug: VRG50635
- Part 2: Cohort 1 VRG50635 (Experimental): Participants will receive VRG50635 (Dose X) for 14 consecutive days.
  Interventions: Drug: VRG50635
- Part 2: Cohort 1 Placebo (Placebo Comparator): Participants will receive VRG50635-matching placebo for 14 consecutive days.
  Interventions: Drug: Placebo
- Part 2: Cohort 2 VRG50635 (Experimental): Participants will receive VRG50635 (Dose Y) for 14 consecutive days.
  Interventions: Drug: VRG50635
- Part 2: Cohort 2 Placebo (Placebo Comparator): Participants will receive VRG50635-matching placebo for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VRG50635 — Specified dose on specified days
  Arms: Part 1: VRG50635 Sequence A, B, C; Part 1: VRG50635 Sequence B, A, C; Part 2: Cohort 1 VRG50635; Part 2: Cohort 2 VRG50635
Drug: Placebo — Specified dose on specified days
  Arms: Part 2: Cohort 1 Placebo; Part 2: Cohort 2 Placebo

SUMMARY:
The primary objectives of this study are to investigate the safety and tolerability of VRG50635 and to determine how VRG50635 is absorbed by the body.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, single-center study conducted in 2 parts to evaluate the safety, tolerability, and PK of VRG50635 following single and multiple doses in healthy participants. The study will consist of a screening period, onsite dosing phase(s), and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 19 and ≤ 55 years of age at Screening.
2. Must be willing and able to voluntarily give written informed consent by signing an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form prior to any study-related procedures being performed.
3. Must have a body mass index ≥ 18.5 and ≤ 32 kilogram per square meter (kg/m2) and weigh ≥ 50 kg.
4. Participants of childbearing potential are eligible to participate if they are not pregnant or breastfeeding and agree to use one highly effective and one barrier method of contraception, if sexually active, for the duration of the study through 90 days after the last study drug administration. Participants must not donate eggs for the duration of study through 90 days after the last dose of study drug.
5. Participants capable of producing sperm must agree that they will use one barrier method of contraception and that their partners of childbearing potential will use one highly effective method of contraception for the duration of the study through 90 days after the last study drug administration. Participants must not donate sperm for the duration of study through 90 days after the last dose of study drug.

Exclusion Criteria:

1. Have a history of clinically significant hematologic, renal, neurologic, pancreatic, gastrointestinal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, immunological, allergic disease, or other major disorders, as determined by the PI.
2. Have any surgical or medical condition that could possibly affect drug absorption (including inflammatory bowel disease, history of gastrectomy, cholecystectomy, or other gastrointestinal tract surgery except appendectomy).
3. Have a current significant medical or psychiatric condition, as determined by the PI.
4. Have a history of serious adverse reaction or serious hypersensitivity to any drug.
5. Have, in the opinion of the PI, evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > the upper limit of normal (ULN) or bilirubin > 1.5 × ULN. Note: Participants with Gilbert syndrome without evidence of hepatic impairment may be enrolled.
6. Have a history or presence of an abnormal electrocardiogram (ECG), including, but not limited to, complete left bundle branch block, second- or third-degree heart block, evidence of prior myocardial infarction, or any other abnormality that is clinically significant in the PI's opinion or precludes accurate interpretation and calculations of cardiac intervals (e.g., QT, QRS).
7. Have clinically significant abnormalities, as assessed by the PI, in laboratory tests at the screening and admission visits. Note: Participants may be rescreened at the discretion of the PI with Sponsor approval.
8. Have abnormal blood pressure: supine systolic blood pressure < 90 or > 140 mmHg, supine diastolic blood pressure < 50 or > 90 mmHg, pulse rate < 40 or > 100 bpm, and body temperature < 35.4 or > 37.8 °C (< 96 or > 100.3 °F) at the screening and admission visits.
9. Have a prolonged corrected QT interval using Fridericia's formula (QTcF) during the 12- lead ECG at Screening or pre-dose on Day 1 > 450 ms for participants assigned male at birth and > 470 ms for participants assigned female at birth.
10. Have a hemoglobin level < 12 g/dL (participants assigned male at birth) or < 10.5 g/dL (participants assigned female at birth).
11. Have participated in any other investigational drug study within 30 days of dosing or within 7 half-lives of the investigational product, whichever is longer, or have previously participated in the current study.
12. Use any prescription medication within 7 days or 5 half-lives (whichever is longer) of the first dose administration and/or anticipated use through the follow-up visit.
13. Use any over-the-counter medication (including vitamin/mineral supplements and herbal medicines, such as St. John's wort and non-standard herbal teas) within 7 days of the first dose administration and/or anticipate using through study participation and the follow-up visit.
14. Receive a positive result in a SARS-CoV-2 test or a COVID-19 vaccine within 30 days prior to Screening.
15. Have poor peripheral venous access.
16. Have donated blood or plasma or otherwise lost ≥ 500 mL of blood within 8 weeks of Screening.
17. Have consumed alcohol, caffeine, or cytochrome P450 (CYP)-altering foods within 48 hours prior to dosing.
18. Have an average daily caffeine intake > 800 mg/day (equivalent to approximately 8 cups of coffee per day).
19. Have a documented medical history of alcoholism or current use of more than 21 units of alcohol per week, of drug abuse, or of drug addiction in the last 2 years.
20. Have a positive drug or alcohol test at Screening.
21. Use tobacco or nicotine products (including tobacco- or nicotine-containing products in any form, including e-cigarettes and vaping) within 90 days before Screening or have a positive nicotine test at the screening or admission visit.
22. Have a history of suicidal behavior or suicidal ideation within the past 60 months, as determined by a positive response ("Yes") to either question 4 or question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening.
23. Have one or more of the following laboratory test abnormalities at Screening: (a) Positive hepatitis C virus (HCV) antibodies; (b) Positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb); (c) Positive HIV 1/2 antibodies.
24. Engage in strenuous activity (including exercise) for ≥ 1 hour within 48 hours of any study day.
25. Are part of the clinical staff personnel or have family members of the clinical site staff or the Sponsor.
26. Have any other issue which, in the opinion of the PI, will make the participant ineligible for study participation.
27. Multiple Dose Part only: Are not eligible for lumbar puncture (have anticoagulation, antiaggregation, or blood coagulation pathologies, history of lumbar spine surgery, acquired or congenital spine malformation, clinical signs of intracranial hypertension, cutaneous infection at the puncture site).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Day 30
Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUCinf) | Up to Day 16
Area Under the Concentration-time Curve from Time 0 to the Last Measurable Concentration (AUClast) | Up to Day 16
Area Under the Concentration-time Curve from Time 0 to 24 Hours Post-dose (AUC0-24) | Up to Day 16
Area Under the Concentration-time Curve Between Consecutive Doses (AUCtau) | Up to Day 16
Maximum Observed Concentration (Cmax) | Up to Day 16
Half-life (t1/2) | Up to Day 16
Time of Maximal Plasma Concentration (tmax) | Up to Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cadavid, MD, Study Director — Verge Genomics
Locations (1):
- Lincoln Celerion Inc.,, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung ST, Linares GR, Chang WH, Eoh Y, Krishnan G, Mendonca S, Hong S, Shi Y, Santana M, Kueth C, Macklin-Isquierdo S, Perry S, Duhaime S, Maios C, Chang J, Perez J, Couto A, Lai J, Li Y, Alworth SV, Hendricks E, Wang Y, Zlokovic BV, Dickman DK, Parker JA, Zarnescu DC, Gao FB, Ichida JK. PIKFYVE inhibition mitigates disease in models of diverse forms of ALS. Cell. 2023 Feb 16;186(4):786-802.e28. doi: 10.1016/j.cell.2023.01.005. Epub 2023 Feb 7. PMID 36754049
- [Background] Shi Y, Lin S, Staats KA, Li Y, Chang WH, Hung ST, Hendricks E, Linares GR, Wang Y, Son EY, Wen X, Kisler K, Wilkinson B, Menendez L, Sugawara T, Woolwine P, Huang M, Cowan MJ, Ge B, Koutsodendris N, Sandor KP, Komberg J, Vangoor VR, Senthilkumar K, Hennes V, Seah C, Nelson AR, Cheng TY, Lee SJ, August PR, Chen JA, Wisniewski N, Hanson-Smith V, Belgard TG, Zhang A, Coba M, Grunseich C, Ward ME, van den Berg LH, Pasterkamp RJ, Trotti D, Zlokovic BV, Ichida JK. Haploinsufficiency leads to neurodegeneration in C9ORF72 ALS/FTD human induced motor neurons. Nat Med. 2018 Mar;24(3):313-325. doi: 10.1038/nm.4490. Epub 2018 Feb 5. PMID 29400714